CLINICAL TRIAL: NCT03237130
Title: Prediction of Lymphatic Metastasis in Esophageal Cancer by CT Radiomics
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Sun Ying-Shi, Chairman of Dept.Radiology of Beijing Cancer Hospital, Peking University Cancer Hospital & Institute
Other Study IDs: CTRadiomics-LMesophagus-BNSF
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Esophagus Cancer
Keywords: esophagus cancer; radiomics; computed tomograpy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative enhanced chest CT: The cohort contains patients with preoperative therapies and patients without preoperative therapies. Each patient receives regular preoperative enhanced chest CT; for patients with preoperative therapies, they usually undergo twice enhanced chest CT examination at before and after preoperative therapies, the CT images after preoperative therapies will be used for analysis
  Interventions: Procedure: preoperative enhanced chest CT examination

INTERVENTIONS:
Procedure: preoperative enhanced chest CT examination — Each patient will receive preoperative enhanced chest CT examination, and their CT images will be used for analysis

SUMMARY:
This study proposes to establish a CT radiomics-based prediction model for identifying metastasis lymph nodes in esophageal cancer.

DETAILED DESCRIPTION:
This study proposes to establish an image feature extraction and selection method for identifying lymph node metastasis of esophageal cancer.The study will consider the relationship between the main lesion and the suspected lymph node, extract association characteristics in order to improve the sensitivity and specificity of the CT radiomics-based prediction model for identifying metastasis lymph nodes. The study includes the construction of CT radiomics-based prediction model and the validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven esophageal cancer
* scheduled to preoperative enhanced chest CT and undergo surgery
* sign the patient informed consent

Exclusion Criteria:

* failed to receive preoperative enhanced chest CT or undergo surgery
* inavailable pathological results for local lymph node status
* inquality of CT images for feature extraction
* patient quit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pathologically proven esophageal cancer patients who receive preoperative CT and surgical resection in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
pathological local lymph node status | Pathologic evaluation will be performed for each patient within 1 week after surgery
  pathological lymph node status is defined as lymph node metastasis exist or not

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, MD, Study Chair — Dept.Radiology,Peking University Cancer Hospital
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided